CLINICAL TRIAL: NCT00903877
Title: T3 for Fibromyalgia: a Pilot Double-blind Non-randomized Clinical Trial
Brief Title: Study of T3 for the Treatment of Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sean Mackey, Assistant Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU-04272009-2419; 16295
Record Dates: First submitted 2009-05-15; First posted 2009-05-19 (Estimated); Results first posted 2017-07-14 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-06

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Triiodothyronine

ARMS (1):
- Placebo followed by T3 (Experimental): Participants receive placebo for 4 weeks. Following placebo, participants begin T3 treatment at 25 mcg per day, for 4 weeks. Following this, participants begin T3 treatment at 50 mcg per day, for 4 more weeks.
  Interventions: Drug: T3

INTERVENTIONS:
Drug: T3 — Patients receive T3 in a dose of 25mcg and 50mcg

SUMMARY:
Determine if T3 - the active form of thyroid hormone - is beneficial in fibromyalgia. Determine the feasibility and promise of an appropriately powered future prospective randomized controlled study of using T3 (the active form of thyroid hormone) for the treatment of fibromyalgia. We specifically aim to assess the feasibility, cost, obstacles and promise of conducting a prospective controlled study in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-50
2. Meet american college of rheumatology criteria for fibromyalgia
3. at baseline report an average pain of 4 or more on a brief Pain Inventory.
4. can climb 2 flights of stairs without shortness of breath.

Exclusion Criteria:

1. new medication change in the last 2 months
2. any cardiac disease at all
3. known thyroid disease before or after thyroid screening bloodwork
4. unstable medical or psychiatric disease.
5. Known inflammatory or rheumatic disease other than fibromyalgia
6. substance abuse in the last year
7. suicidality or depression as indicated by a Beck Depression Inventory of 30 or above
8. concomitant herbal medications
9. multiple severe medication allergies
10. the assessment of the research team that inclusion of the subject could in some way compromise the safety and validity of the study.
11. diabetes
12. smoking
13. Known uncontrolled hypertension
14. known uncontrolled hypercholesterolemia

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2009-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian R Carroll, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo Followed by T3
Started | 51
Completed | 8
Not Completed | 43
Not completed — Did not meet study criteria | 33
Not completed — Withdrawal by Subject | 3
Not completed — Adverse Event | 2
Not completed — Lost to Follow-up | 1
Not completed — Participation put on hold | 4

BASELINE CHARACTERISTICS:
Population: Each participant received placebo followed by 25 mcg of T3.
Arm/Group | Placebo Followed by T3
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 51
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.35 (7.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale of Pain Intensity
Description: Patients rated their pain at baseline, placebo, T3 at 25 mcg, and T3 at 50 mcg. The scale ranged from 0 (no pain) to 10 (pain as bad as it can be).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo Followed by T3
Number analyzed (Participants) | 8
Units on a scale
  Baseline | 6.75 (2.17)
  Placebo | 5.71 (1.82)
  T3 Treatment (25 mcg) | 5.13 (2.95)
  T3 Treatment (50 mcg) | 6.19 (2.37)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the 12 week course of the study.
Description: The clinicaltrials.gov definition of adverse event was used. Adverse events were monitored without regard to the specific Adverse Event Term.
Groups:
- Placebo Followed by T3: All participants receive placebo, followed by 25 mcg of T3.
Arm/Group | Placebo Followed by T3
All-Cause Mortality (participants affected / at risk) | 0/51
Serious Adverse Events (participants affected / at risk) | 1/51
Other Adverse Events (participants affected / at risk) | 1/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Followed by T3 (N=51)
Tachycardia (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Followed by T3 (N=51)
General (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No